CLINICAL TRIAL: NCT00463008
Title: A Pharmacokinetic Study of Methotrexate Using an Intratumoral Microdialysis Catheter
Brief Title: Pharmacologic Study of Methotrexate in Patients Undergoing Stereotactic Biopsy for Recurrent High-Grade Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000346432; NABTT-0302; JHOC-NABTT-0302
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2008-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; recurrent adult brain tumor; adult gliosarcoma; adult giant cell glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — Methotrexate

INTERVENTIONS:
Drug: methotrexate
Other: pharmacological study

SUMMARY:
RATIONALE: Collecting fluid from a brain tumor using a small catheter may help doctors learn how much methotrexate gets into the tumor to kill the tumor cells. It may also help doctors learn how methotrexate works in the brain and in the rest of the body.

PURPOSE: This clinical trial is studying how much methotrexate gets into the brain tumor by collecting fluid directly from the tumor through a small catheter in patients undergoing stereotactic biopsy for recurrent high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of using microdialysis to study distribution of systemically administered methotrexate in the interstitial fluid within a tumor in patients undergoing stereotactic biopsy for recurrent high-grade gliomas.
* Determine the systemic and intratumoral pharmacokinetics of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients have an intratumoral microdialysis catheter placed while undergoing stereotactic biopsy. Between 18-32 hours after placement of catheter, patients receive methotrexate IV over 4 hours. Microdialysis perfusate and blood specimens are collected before, during, and for 24 hours after methotrexate administration.

Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial grade III or IV astrocytoma of 1 of the following subtypes:

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Measurable, contrast-enhancing, residual disease by MRI or CT scan
* Undergoing stereotactic biopsy for confirmation of tumor progression or differentiation of tumor progression from treatment-induced effects

  * Patients with prior low-grade glioma that progressed after prior radiotherapy with or without chemotherapy and in need of stereotactic biopsy to confirm high-grade glioma are eligible
* Must have received prior radiotherapy with or without chemotherapy
* Planning to continue methotrexate therapy after participation on this study
* No ascites or pleural effusions

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 2.0 mg/dL
* SGOT ≤ 4 times upper limit of normal
* Creatinine ≤ 2 mg/dL
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ
* Able to achieve hydration necessary for the use of methotrexate
* Mini mental state exam score at least 15
* No allergy to methotrexate
* No other concurrent infection or medical illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 3 months since prior radiotherapy
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 1 week since prior salicylates, nonsteroidal anti-inflammatory drugs, or sulfonamides
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)
* No concurrent chemotherapeutic agents
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2004-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Comparison of methotrexate levels in the brain extracelluar fluid vs in the serum
Safety and efficacy of the microdialysis catheter

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Olson, MD, Study Chair — Emory University; Stuart A. Grossman, MD — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins